CLINICAL TRIAL: NCT04183764
Title: A Phase Ⅰ Study for Safety, Tolerance, Pharmacokinetic Characteristic of MAX-40279-01 in Patients With Advanced Solid Tumors
Brief Title: MAX-40279-01 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-003
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor
Keywords: advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAX-40279-01 (Experimental): capsule, 5mg and 25mg
  Interventions: Drug: MAX-40279-01

INTERVENTIONS:
Drug: MAX-40279-01 — Part 1: Dose escalation, MAX-40279-01 twice daily with dose modifications based on tolerability criteria.
  Part 2: Dose expansion, Recommended doses from Part 1.

SUMMARY:
This is a multi-center, non-randomized, open-label, single-arm, dose-escalation Phase I study to evaluate the safety and tolerability of MAX-40279-01 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is a two-part study comprised of a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females over age 18.
* Histologically or cytologically confirmed advanced or metastatic solid tumor for which no established standard therapy is available.
* At least one measurable lesion by CT or MRI according to RECIST1.1, which is not in irradiated area (only for expansion phase).
* Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less (in case of alopecia, Grade 2 is acceptable).
* Life expectancy of at least 3 months.
* Female participants of child bearing potential agree not to be pregnant or lactating during the study and for three months following the last dose of study drug. Both men and women of reproductive potential must agree to use a highly effective method of birth control during the study and for three months following the last dose of study drug. A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly.

Exclusion Criteria:

* Any anti-tumor treatment with radiation therapy, surgery, or immunotherapy wihtin 2 weeks (3 weeks for chemotherapy; 6 weeks for nitrosoureas or Mitomycin C) prior to trial entry.
* Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
* Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 2 years at the trial entry.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery.
* Laboratory values not within the Protocol-defined range.
* Cardiac disease , including congestive heart failure, myocardial infarction, unstable arrhythmia, or symptomatic peripheral arterial vascular disease.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD） | 4 weeks
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing.
Adverse events (AEs) | 8 weeks
  Incidence of treatment-related AEs
Phase II dose (RP2D) | 4 weeks
  The number and proportion of patients experiencing at least 1 dose-limiting toxicity (DLT) will be used as the primary measure to evaluate the RP2D of MAX-40279-01.

SECONDARY OUTCOMES:
Tmax | Approximately 4 weeks
  Time to maximum plasma concentration
Cmax | Approximately 4 weeks
  Time to maximum plasma concentration
Objective response rate (ORR) | 12 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No